CLINICAL TRIAL: NCT01434667
Title: Risk Evaluation and Education for Alzheimer's Disease (REVEAL) IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH); University of Michigan (Other); University of Pennsylvania (Other); Howard University (Other)
Responsible Party: Principal Investigator, Robert C. Green, MD, MPH, Principal Investigator, The REVEAL Study, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01HG002213 (NIH); R01HG002213 (NIH)
Record Dates: First submitted 2011-09-07; First posted 2011-09-15 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-09

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment (MCI); Alzheimer's disease (AD); APOE; genetics; risk assessment; education; genetic counseling; Mild Cognitive Impairment, So Stated
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- APOE Genotype Non-Disclosure (Active Comparator): Subjects will receive Alzheimer's disease risk disclosure. This assessment is based on age and MCI status alone.
  Interventions: Behavioral: Alzheimer's disease risk disclosure
- APOE Genotype Disclosure (Experimental): Subjects will receive both APOE genotype and Alzheimer's disease risk disclosure. The assessment is based on age, MCI status, and genotype.
  Interventions: Behavioral: APOE genotype and Alzheimer's disease risk disclosure

INTERVENTIONS:
Behavioral: APOE genotype and Alzheimer's disease risk disclosure — Subjects with MCI will learn their own APOE genotype and a three-year numerical risk estimate for the chance of progressing to dementia of the Alzheimer's type.
  Arms: APOE Genotype Disclosure
Behavioral: Alzheimer's disease risk disclosure — Subjects with MCI will learn a three-year numerical risk estimate for the chance of progressing to dementia of the Alzheimer's type.
  Arms: APOE Genotype Non-Disclosure

SUMMARY:
This study is intended to examine the impact of receiving a genetic risk assessment for Alzheimer's disease (AD) among individuals with Mild Cognitive Impairment (MCI).

DETAILED DESCRIPTION:
Alzheimer's disease is a common condition affecting memory and thinking. Genes can sometimes be used to provide risk estimates for the eventual development of certain common diseases. Apolipoprotein E (APOE) is one gene which can provide information about a person's chances of developing Alzheimer's disease.

Some people with a diagnosis of Mild Cognitive Impairment (MCI) are curious to learn more about the chance of developing Alzheimer's disease. In the REVEAL IV Study, we are examining the psychological and behavioral impact of learning genetic risk information pertaining to the chance for an individual with MCI to progress to dementia of the Alzheimer's type within three years.

Participation in this study requires an initial phone call which will elicit some demographic information about the participant and his or her study partner. A first in-person visit to the research clinic will consist of an education session, the administration of knowledge and attitudinal surveys and some tests to assess memory and thinking skills. This visit will take approximately 2-3 hours. Participants with MCI will have their blood drawn for genetic testing. Participants will then be randomized to one of two groups. Those in the intervention arm will receive a three-year risk estimate for the chance of progressing to dementia of the Alzheimer's type based on age, the diagnosis of MCI and their own APOE gene test result. Those in the comparison arm will receive a three-year risk estimate for the chance of progressing to dementia of the Alzheimer's type based on age and the diagnosis of MCI, without the APOE gene test result. Participants randomized to the comparison arm will have the opportunity to learn their own APOE gene test result at the end of the study. Participants and their study partners will be followed for 6 months following disclosure of results with 1 additional clinic visit and 1 additional phone interviews.

ELIGIBILITY:
Inclusion Criteria:

* Individuals (55-90 years old) with Mild Cognitive Impairment (amnestic-MCI as defined by the Petersen criteria)
* Individuals who have a close friend, relative or spouse (18+) willing to be a study partner. Study partners attend each study visit with the participant and also complete surveys and interviews.

Exclusion Criteria:

* Individuals with current, untreated anxiety or depression
* Individuals who do not meet the criteria for amnestic-MCI
* Individuals who have the diagnosis of dementia or Alzheimer's disease
* Individuals not fluent in English
* Individuals who do not have a study partner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2010-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Green, MD, MPH, Principal Investigator — Brigham and Women's Hospital/Harvard Medical School
Locations (3):
- United States (3):
  - Howard University, Washington D.C., District of Columbia
  - University of Michigan, Ann Arbor, Michigan
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Roberts JS, Karlawish JH, Uhlmann WR, Petersen RC, Green RC. Mild cognitive impairment in clinical care: a survey of American Academy of Neurology members. Neurology. 2010 Aug 3;75(5):425-31. doi: 10.1212/WNL.0b013e3181eb5872. PMID 20679636
- [Background] Roberts JS, Christensen KD, Green RC. Using Alzheimer's disease as a model for genetic risk disclosure: implications for personal genomics. Clin Genet. 2011 Nov;80(5):407-14. doi: 10.1111/j.1399-0004.2011.01739.x. Epub 2011 Jul 18. PMID 21696382
- [Result] Guan Y, Roter DL, Wolff JL, Gitlin LN, Christensen KD, Roberts JS, Green RC, Erby LH. The impact of genetic counselors' use of facilitative strategies on cognitive and emotional processing of genetic risk disclosure for Alzheimer's disease. Patient Educ Couns. 2018 May;101(5):817-823. doi: 10.1016/j.pec.2017.11.019. Epub 2017 Nov 27. PMID 29203084
- [Result] Guan Y, Roter DL, Erby LH, Wolff JL, Gitlin LN, Roberts JS, Green RC, Christensen KD. Disclosing genetic risk of Alzheimer's disease to cognitively impaired patients and visit companions: Findings from the REVEAL Study. Patient Educ Couns. 2017 May;100(5):927-935. doi: 10.1016/j.pec.2016.12.005. Epub 2016 Dec 14. PMID 28012682
- See also: Alzheimer's Association - Educational Materials on Mild Cognitive Impairment — https://www.alz.org/alzheimers-dementia/what-is-dementia/related_conditions/mild-cognitive-impairment
- See also: Alzheimer's Association - Educational Materials on Risk Factors — http://www.alz.org/alzheimers_disease_causes_risk_factors.asp
- See also: REVEAL Study overview — http://www.genomes2people.org/research/reveal/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 32 enrolled participants were not assigned for the reasons that follow:
  Ineligible (n=7)
  * No study partner: 5
  * Diagnosis was not amnestic mild cognitive impairment (MCI): 1
  * Low cognitive score: 1
  Declined to continue (n=17)
  * No longer interested: n=11
  * Too busy: 4
  * No reason given: 2
  Lost to follow-up (n=8)
Groups:
- Apolipoprotein E (APOE) Genotype Non-Disclosure: Subjects will receive Alzheimer's disease risk disclosure. This assessment is based on age and MCI status alone.
  Alzheimer's disease risk disclosure: Subjects with MCI will learn a three-year numerical risk estimate for the chance of progressing to dementia of the Alzheimer's type.
- Apolipoprotein E (APOE) Genotype Disclosure: Subjects will receive both APOE genotype and Alzheimer's disease risk disclosure. The assessment is based on age, MCI status, and genotype.
  APOE genotype and Alzheimer's disease risk disclosure: Subjects with MCI will learn their own APOE genotype and a three-year numerical risk estimate for the chance of progressing to dementia of the Alzheimer's type.
Period: Overall Study
Arm/Group | Apolipoprotein E (APOE) Genotype Non-Disclosure | Apolipoprotein E (APOE) Genotype Disclosure
Started | 39 | 75
Completed | 34 | 65
Not Completed | 5 | 10
Not completed — Lost to Follow-up | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | APOE Genotype Non-Disclosure | APOE Genotype Disclosure | Total
Number analyzed (Participants) | 39 | 75 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 11 | 14
  >=65 years | 36 | 64 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.1 (8.1) | 73.3 (7.3) | 73.9 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 39 | 57
  Male | 21 | 36 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 36 | 72 | 108
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Self-identified race
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 9 | 11 | 20
    White | 30 | 64 | 94
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 75 | 125

OUTCOME MEASURES:

1. Primary Outcome: Geriatric Depression Scale
Description: A 15-item self-report assessment used to identify depression in the elderly. GDS scores ranged from 0-15. Higher scores indicated greater depression.
Time Frame: Baseline, 6 weeks post-disclosure, and 6 months post-disclosure
Population: Participants who completed the full 15-item scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | APOE Genotype Non-Disclosure | APOE Genotype Disclosure
Number analyzed (Participants) | 39 | 75
score on a scale
  Baseline | 2.6 (2.6) | 2.1 (2.0)
  6 Weeks Post-Disclosure: number analyzed (Participants) | 37 | 74
  6 Weeks Post-Disclosure | 2.8 (2.7) | 1.9 (1.6)
  6 Months Post-Disclosure: number analyzed (Participants) | 34 | 64
  6 Months Post-Disclosure | 2.1 (2.2) | 2.0 (2.1)

2. Primary Outcome: Mini State Trait Anxiety Inventory
Description: Validated introspective psychological inventory consisting of 6 self-report items pertaining to anxiety affect. Responses are transformed into scores that range from 20 to 80, with higher scores indicating greater anxiety.
Time Frame: Baseline, 6 weeks post-disclosure, and 6 months post-disclosure
Population: Participants who completed the full 6-item scale
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | APOE Genotype Non-Disclosure | APOE Genotype Disclosure
Number analyzed (Participants) | 39 | 75
score on a scale
  Baseline | 36.3 (12.0) | 36.5 (10.9)
  6 Weeks Post-Disclosure: number analyzed (Participants) | 37 | 74
  6 Weeks Post-Disclosure | 39.0 (13.6) | 36.6 (11.8)
  6 Months Post-Disclosure: number analyzed (Participants) | 34 | 65
  6 Months Post-Disclosure | 36.2 (12.3) | 36.2 (13.4)

3. Secondary Outcome: Impact of Event Scale (IES)
Description: The Impact of Event assesses intrusive thoughts and avoidance related to a specific stressful life event. It is a 15-item self-report measure with scores that range from 0 to 75, with greater scores indicating greater distress about the event.
Time Frame: 1-3 Days, 6 Weeks and 6 Months Post-disclosure
Population: Participants who completed the full 15-item scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | APOE Genotype Non-Disclosure | APOE Genotype Disclosure
Number analyzed (Participants) | 37 | 74
score on a scale
  1-3 Days Post-Disclosure | 8.2 (8.7) | 8.1 (9.4)
  6 Weeks Post-Disclosure: number analyzed (Participants) | 36 | 74
  6 Weeks Post-Disclosure | 13.1 (11.4) | 11.5 (12.6)
  6 Months Post-Disclosure: number analyzed (Participants) | 33 | 65
  6 Months Post-Disclosure | 12.5 (11.9) | 12.4 (12.0)

4. Secondary Outcome: Psychological Impact of Test Disclosure (IGT-AD)
Description: A 15-item scale measuring distress specific to the test results received. Scores range from 0-75, with higher scores indicating greater test-related distress. Higher scores indicate greater distress about the risk assessment.
Time Frame: 6 Weeks and 6 Months Post-disclosure
Population: Participants who completed the full 15-item scale
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | APOE Genotype Non-Disclosure | APOE Genotype Disclosure
Number analyzed (Participants) | 34 | 73
score on a scale
  6 Weeks Post-Disclosure | 24.7 (10.0) | 19.5 (11.5)
  6 Months Post-Disclosure: number analyzed (Participants) | 30 | 64
  6 Months Post-Disclosure | 24.1 (10.8) | 20.3 (11.2)

5. Secondary Outcome: Recall and Comprehension of Risk Information
Description: Several measures to assess participant recall and comprehension of personalized risk information for AD. The sum number correct of the two items that were presented to both randomization arms ("What form of APOE increases risk for Alzheimer's disease?", and "What percentage were you given as your 3-year risk of developing Alzheimer's disease?") are summarized here.
Time Frame: 6 Weeks and 6 Months Post-disclosure
Population: Participants who provided data on each scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | APOE Genotype Non-Disclosure | APOE Genotype Disclosure
Number analyzed (Participants) | 34 | 63
score on a scale
  6 Weeks Post-Disclosure | 0.8 (0.7) | 1.2 (0.8)
  6 Months Post-Disclosure: number analyzed (Participants) | 26 | 52
  6 Months Post-Disclosure | 1.0 (0.7) | 1.2 (0.7)

6. Secondary Outcome: Participant Satisfaction
Description: How well participants' expectations about information, explanations, reassurance, advice, and help in decision making were met. Participants rated satisfaction for each dimension on a 1-7 scale, with higher scores indicating that expectations were met better.
Time Frame: 6 Weeks and 6 Months Post-disclosure
Population: Participants who provided responses on each expectation item
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | APOE Genotype Non-Disclosure | APOE Genotype Disclosure
Number analyzed (Participants) | 37 | 73
score on a scale
  Information: 6 Weeks Post-Disclosure | 6.0 (1.1) | 6.1 (1.2)
  Explanation: 6 Weeks Post-Disclosure: number analyzed (Participants) | 37 | 71
  Explanation: 6 Weeks Post-Disclosure | 5.9 (1.2) | 6.2 (1.2)
  Reassurance: 6 Weeks Post-Disclosure: number analyzed (Participants) | 35 | 70
  Reassurance: 6 Weeks Post-Disclosure | 5.5 (1.5) | 6.0 (1.3)
  Advice: 6 Weeks Post-Disclosure: number analyzed (Participants) | 35 | 70
  Advice: 6 Weeks Post-Disclosure | 5.6 (1.4) | 5.4 (1.7)
  Help in decision making: 6 Weeks Post-Disclosure: number analyzed (Participants) | 35 | 71
  Help in decision making: 6 Weeks Post-Disclosure | 5.2 (1.7) | 5.3 (1.6)
  Information: 6 Months Post-Disclosure: number analyzed (Participants) | 30 | 62
  Information: 6 Months Post-Disclosure | 5.6 (1.4) | 6.1 (1.2)
  Explanation: 6 Months Post-Disclosure: number analyzed (Participants) | 30 | 62
  Explanation: 6 Months Post-Disclosure | 5.7 (1.3) | 6.2 (1.0)
  Reassurance: 6 Months Post-Disclosure: number analyzed (Participants) | 30 | 62
  Reassurance: 6 Months Post-Disclosure | 5.5 (1.2) | 5.8 (1.3)
  Advice: 6 Months Post-Disclosure: number analyzed (Participants) | 30 | 61
  Advice: 6 Months Post-Disclosure | 5.4 (1.3) | 5.6 (1.4)
  Help in decision making: 6 Months Post-Disclosure: number analyzed (Participants) | 30 | 60
  Help in decision making: 6 Months Post-Disclosure | 5.2 (1.3) | 5.6 (1.4)

7. Secondary Outcome: User Ratings of Risk Assessment Experience
Description: Subjective ratings of the impact of risk assessment. Participants provided ratings on a 1-5 scale, with 1 being "very negative" and 5 being "very positive"
Time Frame: 6 Weeks and 6 Months Post-disclosure
Population: Participants who completed these items in the post-disclosure surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | APOE Genotype Non-Disclosure | APOE Genotype Disclosure
Number analyzed (Participants) | 35 | 73
score on a scale
  6 Weeks Post-Disclosure | 3.5 (0.9) | 3.6 (1.0)
  6 Months Post-Disclosure: number analyzed (Participants) | 31 | 65
  6 Months Post-Disclosure | 3.0 (0.8) | 3.5 (1.0)

8. Secondary Outcome: Health Behavior and Insurance Changes
Description: AD prevention behaviors enacted within the prior two weeks.
Time Frame: Baseline, 6 weeks post-disclosure, and 6 months post-disclosure
Population: Participants who provided data on health behaviors at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | APOE Genotype Non-Disclosure | APOE Genotype Disclosure
Number analyzed (Participants) | 39 | 75
Participants
  Baseline: Diet | 6 | 17
  Baseline: Physical activity | 16 | 26
  Baseline: Dietary supplements | 7 | 15
  Baseline: Mental activities | 13 | 37
  Baseline: Stress management | 1 | 10
  Baseline: Medications | 8 | 26
  6 Weeks post-disclosure: Diet: number analyzed (Participants) | 38 | 74
  6 Weeks post-disclosure: Diet | 9 | 16
  6 Weeks post-disclosure: Physical activity: number analyzed (Participants) | 38 | 74
  6 Weeks post-disclosure: Physical activity | 16 | 30
  6 Weeks post-disclosure: Dietary supplements: number analyzed (Participants) | 38 | 74
  6 Weeks post-disclosure: Dietary supplements | 9 | 25
  6 Weeks post-disclosure: Mental activities: number analyzed (Participants) | 38 | 74
  6 Weeks post-disclosure: Mental activities | 12 | 38
  6 Weeks post-disclosure: Stress management: number analyzed (Participants) | 38 | 74
  6 Weeks post-disclosure: Stress management | 6 | 20
  6 Weeks post-disclosure: Medications: number analyzed (Participants) | 38 | 74
  6 Weeks post-disclosure: Medications | 7 | 24
  6 Months post-disclosure: Diet: number analyzed (Participants) | 31 | 63
  6 Months post-disclosure: Diet | 6 | 20
  6 Months post-disclosure: Physical activity: number analyzed (Participants) | 31 | 63
  6 Months post-disclosure: Physical activity | 12 | 23
  6 Months post-disclosure: Dietary supplements: number analyzed (Participants) | 31 | 63
  6 Months post-disclosure: Dietary supplements | 9 | 16
  6 Months post-disclosure: Mental activities: number analyzed (Participants) | 31 | 65
  6 Months post-disclosure: Mental activities | 15 | 40
  6 Months post-disclosure: Stress management: number analyzed (Participants) | 32 | 63
  6 Months post-disclosure: Stress management | 3 | 18
  6 Months post-disclosure: Medications: number analyzed (Participants) | 31 | 64
  6 Months post-disclosure: Medications | 4 | 22

9. Secondary Outcome: Insurance and Advance Planning Changes
Description: A series of yes/no questions that ask whether the risk assessment motivated changes to insurance or advance planning.
Time Frame: 6 months post-disclosure
Population: Participants who provided data on the 6-month follow-up survey about these outcomes
Measure: Count of Participants; unit: Participants
Arm/Group | APOE Genotype Non-Disclosure | APOE Genotype Disclosure
Number analyzed (Participants) | 31 | 64
Participants
  Health insurance change | 2 | 1
  Life insurance change | 0 | 1
  Short-term disability insurance change | 0 | 0
  Long-term disability insurance | 0 | 0
  Long-term care insurance | 0 | 0
  Change to will: number analyzed (Participants) | 28 | 54
  Change to will | 0 | 0
  Change to living will: number analyzed (Participants) | 25 | 51
  Change to living will | 1 | 1
  Change to durable power of attorney: number analyzed (Participants) | 21 | 50
  Change to durable power of attorney | 0 | 0

10. Secondary Outcome: Participation in Alzheimer's Disease-related Research After Receiving the Alzheimer's Disease Risk Estimate.
Description: Yes/no response to the question, "Since receiving your Alzheimer's disease risk estimate, have you joined any other Alzheimer's disease-related research studies?"
Time Frame: 6 weeks and 6 months post-disclosure
Population: Participants who provided data on these survey items
Measure: Count of Participants; unit: Participants
Arm/Group | APOE Genotype Non-Disclosure | APOE Genotype Disclosure
Number analyzed (Participants) | 37 | 74
Participants
  6 Weeks post-disclosure | 0 | 6
  6 Months post-disclosure: number analyzed (Participants) | 33 | 66
  6 Months post-disclosure | 2 | 10

ADVERSE EVENTS:
Time Frame: From enrollment through 6 months after the Alzheimer's disease risk assessment.
Description: Non-serious adverse events were defined as scores at any time including baseline, on psychological outcome scales greater than or equal to 56 on the STAI (anxiety), 8 on the GDS (depression) or 2 on the BHS (hopelessness). Non-serious adverse events were identified at the judgment of study personnel as events that caused inconvenience or concern to participants, but did not qualify as serious. Serious adverse events were defined per guidelines from the National Institutes of Aging.
Arm/Group | APOE Genotype Non-Disclosure | APOE Genotype Disclosure
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/75
Other Adverse Events (participants affected / at risk) | 16/39 | 18/75
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | APOE Genotype Non-Disclosure (N=39) | APOE Genotype Disclosure (N=75)
Increased monitoring due to high scores on anxiety, depression or hopelessness scales (Psychiatric disorders) | 16 | 17 — Scores at any time point of 56 or higher on the 6-item State-Trait Anxiety Index (STAI), 8 or higher on the 15-item Geriatric Depression Scale (GDS), and 2 or higher on the 4-item Beck Hopelessness Scale (BHS).
Delayed disclosure session (Investigations) | 0 | 1 — Extended delay of disclosure of Alzheimer's disease risk assessment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No